CLINICAL TRIAL: NCT02321358
Title: Randomized Controlled Trial of a Behavior Change Intervention to Increase Aerobic and Resistance Exercise and Quality of Life in Older Prostate and Breast Cancer Survivors: The OutPACE Trial
Brief Title: Trial of a Behavior Change Intervention to Increase Aerobic and Resistance Exercise and Quality of Life in Older Prostate and Breast Cancer Survivors
Acronym: OutPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Collaborators: Mitacs (Industry)
Responsible Party: Principal Investigator, Erin McGowan, Assistant Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20141338-HK
Record Dates: First submitted 2014-12-08; First posted 2014-12-22 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Quality of Life; Physical Activity; Fatigue; Breast Cancer; Prostate Cancer
Keywords: Behavior Change; Objectively Measured Physical Activity; Survivorship
MeSH Terms: conditions — Motor Activity; Fatigue; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Two-time implementation intention (Experimental): Group will receive physical activity materials along with the implementation intention intervention and a booster again six weeks following.
  Interventions: Behavioral: Two-time implementation intention; Behavioral: Physical Activity Materials
- One-time implementation intention (Active Comparator): Group will receive physical activity materials along with the implementation intention intervention.
  Interventions: Behavioral: One-time implementation intention; Behavioral: Physical Activity Materials
- Sham Comparator Group (Sham Comparator): Group will receive Canada's Food Guide which contains a small amount of physical activity information.
  Interventions: Behavioral: Sham Comparator

INTERVENTIONS:
Behavioral: Two-time implementation intention — Will be given intervention and booster at six weeks
  Arms: Two-time implementation intention
Behavioral: One-time implementation intention — Will only be given the intervention once
  Arms: One-time implementation intention
Behavioral: Sham Comparator — Canada's Food Guide for Healthy Eating will be provided. This contains a small amount of physical activity information.
  Arms: Sham Comparator Group
Behavioral: Physical Activity Materials — Thera-Bands, instructional DVD and exercise handout, instructional stretching handout, CSEP Physical activity guidelines.
  Arms: One-time implementation intention; Two-time implementation intention

SUMMARY:
This trial is a three-armed randomized controlled trial which will explore the utility of an implementation intention intervention on aerobic and resistance exercise in older (60+) prostate and breast cancer survivors and improving quality of life. It is expected that those in the experimental groups will report greater increases in their physical activity, resulting in greater improvements in their quality of life.

DETAILED DESCRIPTION:
Recruitment

Potential participants will be contacted by the Newfoundland and Labrador Cancer registry. They will be given a brief explanation of the study will be asked to consent to a mail-out questionnaire from the registry. The questionnaire will contain a cover letter explaining the study in more detail along with informed consent. If the participant wishes to continue in the study, they will return the questionnaire to the research team, who will contact them from this point.

Participants will also be recruited through presentations at local support groups as well as advertisements in local papers and posters at local hospitals and recreation centers.

Power Analysis

According to G*Power a sample of 40 prostate and breast cancer survivors per group (n=120) is needed to detect a medium effect size (d= .50) on our primary outcome (i.e., PA) with a power of 0.80, at a p-level of 0.05. We expect a 20% attrition rate, based on previous research (McGowan, North, & Courneya, 2013; Vallance, Courneya, Plotnikoff, Yasui, & Mackey, 2007) therefore we will attempt to recruit a sample of 150 breast and prostate cancer survivors, which would allow for 50 participants per group.

Data Analysis

Analyses of covariance will be used to examine group differences on our primary outcome (i.e., PA minute/week) at month 1 and month 3, and secondary outcomes (e.g., QoL) at month 3. Additional analyses of covariance will be run to explore the group differences on sedentary behaviour, and light, moderate and vigorous minutes of activity/week at month 1 and month 3. Medical (e.g., comorbidities, months since diagnosis) and demographic (e.g., marital status, age, BMI) will be tested as possible moderators of PA behaviour change.

If we experience a large proportion of missing data multiple imputation techniques in SPSS will be used to replace missing values. Otherwise, a last outcome carried forward approach will be used.

The relationships between self-reported PA and QoL, and objectively measured PA and QoL in older breast and prostate cancer survivors will be explored. To examine this, differences in QoL between participants in the two PA categories (i.e., meeting PA guidelines and not meeting PA guidelines) will be tested using analysis of variance (ANOVA). These analyses will be repeated using analysis of covariance (ANCOVA) to control for the demographic and medical variables that had statistically significant associations with the QoL.

The relationship between objectively measured PA and self-reported PA will be explored using a two-way mixed intraclass correlation coefficient to calculate the level of absolute agreement between the two types of measurements.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or older
* Breast or prostate cancer survivor
* Completed surgery, radiation and/or chemotherapy
* Proficient in English
* Living in the greater St. John's, NL area; participants are asked to meet researchers at the university
* Have an interest in becoming more active or learning about physical activity

Exclusion Criteria:

* Those with contraindications to exercise
* Participants will be asked about other existing diseases and if they have been told by their doctor to avoid certain activities. Some may be asked to consult with physician before taking part

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change in Self-Reported Physical Activity | Baseline, one month follow-up, three month follow-up
  Using Godin's Leisure Score Index, participants will be asked how much physical activity they took part in over the past seven days. Data from each time point will be analyzed and compared to determine change.
Change in Objectively Measured Physical Activity | Baseline, one month follow-up, three month follow-up
  Participants will wear an accelerometer (ActiGraph GT3X) for seven days to assess their activity. Data from each time point will be analyzed and compared to determine change.

SECONDARY OUTCOMES:
Change in Fatigue | Baseline, one month follow-up, three month follow-up
  Will be assessed using the FACIT-F questionnaire. Data from each time point will be analyzed and compared to determine change.
Change in Quality of Life | Baseline, one month follow-up, three month follow-up
  Will be assessed using the short-form 36 scale (SF-36) and Functional Assessment of Cancer Therapy (FACT) questionnaire, specific to cancer type (FACT-Breast or FACT-Prostate). Data from each time point will be analyzed and compared to determine change.

CONTACTS AND LOCATIONS:
Overall Officials: Erin L McGowan, Ph.D, Principal Investigator — Assistant Professor
Locations (1):
- School of Human Kinetics and Recreation, St. John's, Newfoundland and Labrador, Canada

REFERENCES:
- [Background] McGowan EL, North S, Courneya KS. Randomized controlled trial of a behavior change intervention to increase physical activity and quality of life in prostate cancer survivors. Ann Behav Med. 2013 Dec;46(3):382-93. doi: 10.1007/s12160-013-9519-1. PMID 23783829
- [Background] Vallance JK, Courneya KS, Plotnikoff RC, Yasui Y, Mackey JR. Randomized controlled trial of the effects of print materials and step pedometers on physical activity and quality of life in breast cancer survivors. J Clin Oncol. 2007 Jun 10;25(17):2352-9. doi: 10.1200/JCO.2006.07.9988. PMID 17557948